CLINICAL TRIAL: NCT05599880
Title: A Phase 2 Study to Investigate Efficacy and Safety Evaluation of Bortezomib in Patients With Relapsed/Refractory Immune Thrombocytopenia
Brief Title: The Investigate Efficacy and Safety Evaluation of Bortezomib in Patients With Relapsed/Refractory Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong-Yeop Shin, hematology oncology Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BORRELIA
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Bortezomib is administered at 1.3mg/m2 iv or sc on each Cycly Day1, Days4, and Days8. Bortezomib is administered every 3 weeks for a total of 3 cycles. Thereafter, follow-up is scheduled for 12 months.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib is administered at 1.3mg/m2 iv or sc on each Cycly Day1, Days4, and Days8. Bortezomib is administered every 3 weeks for a total of 3 cycles. Thereafter, follow-up is scheduled for 12 months.

SUMMARY:
to investigate efficacy and safety evaluation of bortezomib in patients with relapsed/refractory immune thrombocytopenia

DETAILED DESCRIPTION:
A sufficient explanation of the study should be provided to outpatients or inpatients who meet the research subject selection criteria. Then, it is conducted for those who have given their voluntary consent to participate in the study. Those enrolled in the study conduct according to the criteria specified in the protocol. In this clinical trial, 3 weeks is defined as 1 cycle. A total of 3 cycles will be performed, and follow-up will be conducted for 12 months. The study subjects will receive the test drug on an outpatient basis. At each outpatient visit, vital signs, medical history, physical examination, ECOG evaluation and blood tests are performed, and adverse reactions are checked. Bone marrow blood test is performed as an option at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 19 years of age and older
2. Patients diagnosed with immune thrombocytopenia (primary or secondary)
3. (Patients with at least one of B, C, or D meeting A below.) A.A person who has been confirmed not to be due to a cause of decreased platelet production in the bone marrow in the results of bone marrow examination within the past 5 years. (Bone marrow examination is required if there is no bone marrow examination result within the last 5 years.) B.After being diagnosed with ITP, there has been a case of complete platelet response with plt >100k in immunoglobulin therapy.

   C.Patients suspected of having primary immune thrombocytopenia with proven anti-platelet antibody., D.Helicobacter IgG, antinuclear antibody (ANA), anticardiolipin antibody (ACA), nonspecific inhibitor (NSI), etc. have been proven, and secondary immune thrombocytopenia caused by autoimmune disease is suspected.
4. platelets <30 x 109/L
5. Patients in need of clinical treatment.
6. Patients who have relapsed or refractory after receiving treatment with corticosteroids (prednisolone cumulative dose 5.6mg/kg (0.8mg/kg 1 week) or more or dexamethasone cumulative dose 80mg (20mg 4 days) or more)., However, there are exceptions when corticosteroids are contraindicated.
7. Patients who have been relapsed or refractory after receiving at least 2 treatments with a mechanism other than corticosteroids.
8. Patients who underwent two different treatments from among the treatment methods below.

   * Splenectomy
   * eltrombopag or romiplostim
   * Rituximab treatment
   * Azathioprine
   * cyclosporine or mycophenolate mofetil(MMF)
   * vincristine or cyclophosphamide
   * danazol
   * dapsone
   * Alemtuzumab
9. Female patients of childbearing potential should have a negative urine or serum pregnancy test within 28 days before starting administration of the test drug.
10. Patients who voluntarily or legal guardians have given written consent to participate in this clinical trial.

Exclusion Criteria:

1. pregnant, lactating women
2. Patients allergic to bortezomib.
3. Patients with Grade 2 or higher peripheral neuropathy requiring drug treatment.
4. Patients with severe or uncontrolled active infection.
5. Patients with significant immunoglobulin degradation in the immunoglobulin profile.
6. HBV, HCV carrier or HIV patient. (However, if the patient is being stably maintained with antiviral treatment, and the expert opinion determines that it is possible to participate in the clinical trial along with antiviral treatment and prevention, participation is possible.)
7. Patients currently undergoing chemotherapy.
8. Patients whose bone marrow did not recover after cancer treatment, or whose cause other than immune destruction was confirmed by bone marrow examination, such as thrombocytopenia due to intramedullary abnormalities. However, if the presence of anti-platelet antibodies is proven and thrombocytopenia due to immune destruction is strongly suspected clinically, registration is possible even if there are other causes of thrombocytopenia.)
9. Patients who may become pregnant. However, women of childbearing age(If postmenopausal women are not of childbearing age, they must have been menstruating for at least 12 months.) who have not undergone sterilization can participate in the clinical trial only if the pregnancy test is negative. And, effective contraception must be maintained throughout the entire trial period.
10. Patients currently participating in other clinical trials.
11. Patients who are not considered suitable for participation in clinical trials in the opinion of the researcher.
12. Patients with inadequate organ function.

    * total bilirubin > 3 x ULN
    * creatinine > 1.5 x ULN
    * liver function test AST(SGOT) & ALT(SGPT) > 3 x ULN

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmation of efficacy of bortezomib in patients with relapsed/refractory immune thrombocytopenia requiring treatment | at week 9.
  platelet >30 x 109/L and at least twofold increase from baseline; complete >100 x 109/L, partial 30-100 x 109/L, Platelet response rate at week 9.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Yeop Shin, MD, PhD, Study Chair — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Guri-si
  - Seoul National University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul